CLINICAL TRIAL: NCT05080309
Title: Effect of Oral Carbohydrate Intake > 44kCal Per Hour During Labour on the Rate of Instrumental Vaginal Delivery
Acronym: soliso-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21-0017
Record Dates: First submitted 2021-07-22; First posted 2021-10-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Delivery Complication; Labor Long; Pregnancy Related
Keywords: labor; instrumental vaginal delivery; oral intake; nulliparous

STUDY DESIGN:
Intervention Model Description: controlled and monitored oral fruit juice intake in order to achieve an oral calory intake > 44kCal/hour during labor
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor (i.e. obstetrician) will be unaware of group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Sham Comparator): During labor the women will have free access to water only but not fruit juice or other calory source.
  Interventions: Other: free water only
- Carbohydrate (Experimental): During labor the women will have free access to water and 20 ml commercial fruit juice bricks containing between 430 or 660 kcal/l. Every 2 hours the midwife or the nurse will measure the fruit juice oral intake volume and will advise women to drink the planned volume (1 brick/2hours)
  Interventions: Dietary Supplement: carbohydrate oral intake

INTERVENTIONS:
Dietary Supplement: carbohydrate oral intake — During labor the women will have free access to water and 20 ml commercial fruit juice bricks containing between 430 or 660 kcal/l. Every 2 hours the midwife or the nurse will measure the fruit juice oral intake volume and will advise women to drink the planned volume (1 brick/2hours)
  Arms: Carbohydrate
Other: free water only — Women will have free access to water only
  Arms: Control

SUMMARY:
Carbohydrate intake during physical exercise improves muscle performance and decreases fatigue. We hypothesized that carbohydrate intake during labor which is a period of significant physical activity can decrease the instrumental vaginal delivery rate.

In a previous study we reported a trend toward a decrease in instrumental vaginal delivery and the mount of carbohydrate intake during labour. However due to some limitations no clear conclusion could be drawn.

The present study is designed to examine the relationship between a high calory oral intake (>44 kCal/hour during labour) and the rate of instrumental delivery.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women
* singleton pregnancy
* social insurance
* uncomplicated pregnancy
* no contraindication to vaginal delivery

Exclusion Criteria:

* scheduled caesarean section
* labor < 37 weeks of gestational age
* cervical dilation > 8cm at inclusion
* scheduled induced delivery
* contraindication to pushing effort during labor and delivery
* BMI > 40 kg/m2
* medical history of diabetes mellitus, hypertension, heart disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — nullparous pregnant women during labor and delivery
Enrollment: 600 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-09-03 (Estimated)

PRIMARY OUTCOMES:
instrumental vaginal delivery | 2 days
  rate of instrumental vaginal delivery

SECONDARY OUTCOMES:
oxytocin administration | 2 days
  rate of oxytocin administration
caesarean section | 2 days
  rate of caesarean section
nausea and vomiting | 2 days
  rate of nausea and vomiting
thirst sensation on verbal rating scale | 2 days
  self evaluation of thirst using a verbal rating scale from 0 (not thirst to 10 maximal thirst)
hunger sensation on verbal rating scale | 2 days
  self evaluation of hunger using a verbal rating scale from 0 (no hunger to 10 maximal hunger)
fatigue | 2 days
  self evaluation of fatigue using a verbal rating scale from 0 (0 no fatigue to 10 exhausted)
umbilical blood pH | 1 min
  umbilical blood pH measured at child birth

CONTACTS AND LOCATIONS:
Overall Officials: jean-luc hanouz, M.D., Ph.D., Study Chair — University Hospital of Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No